## Document Cover Page

## Official Title of the Study:

Responsible Fatherhood Opportunities for Reentry & Mobility (ReFORM)

NCT Number: NCT02860988

**Date of Document:** September 29, 2020

# Responsible Fatherhood Opportunities for Reentry & Mobility (ReFORM) Protocol

#### Background

Mountain Comprehensive Care Center (MCCC) in Prestonsburg, KY was recently awarded a grant from the Administration for Children and Families (ACF) as part of the Responsible Fatherhood Opportunities for Reentry and Mobility (ReFORM) Program to strengthen positive father-child engagement, improve employment and economic mobility opportunities, improve healthy relationships and marriage, and decrease barriers to successful community reentry. MCCC has a physical presence in Floyd, Johnson, Lawrence, Magoffin, Martin and Pike in eastern Kentucky and established relationships with the two targeted detention centers for pre-release services (Floyd County Detention Center and Big Sandy Regional Detention Center).

To address barriers to service participation, grant funding will be used to provide evidence-based services to strengthen parenting skills for fathers who are incarcerated and planning for community re-entry, along with interventions to increase economic mobility and relationships. Individualized, culturally- /gender- competent and comprehensive case management and wraparound services will also foster program participation and success. The project will offer integrated services for fathers who are incarcerated in the targeted area who are incarcerated in Floyd County or Big Sandy facilities. Responsible parenting activities will include skills-based parenting education, dissemination of information regarding good parenting practices, one-on-one counseling regarding parenting issues, and will encourage and seek to facilitate the financial support of participants' children. Economic stability activities will include job readiness workshops, and upon release, linkages with additional job training and educational assistance, job search and placement assistance as well as employment incentives at 30 days of employment. Finally, healthy marriage/relationship activities will include marriage and relationship education, conflict resolution skills training, financial literacy seminars and counseling. Semi-annual parent/child events and annual relationship events will also be available to foster stronger family connections.

## **Objectives**

The ACF award to MCCC primarily supports service enhancement and service delivery. To ensure the effectiveness of the proposed services, MCCC will be contracting with University of Kentucky to perform the evaluation. The evaluation includes two primary components:

- consultation on the collection of ACF required Performance Measures to document program client characteristics, program operations, enrollment and participation, and pre-test/post-test outcome measures; and
- 2) responsibility for the local evaluation which includes a quasi-experimental two group design to examine the effectiveness of targeted services for fathers at MCCC

#### Study Design

The local evaluation will utilize a quasi-experimental research design including an experimental group (receives MCCC targeted services under the newly funded ACF grant) and a comparison group (incarcerated fathers who do not receive targeted services in a comparable local regional jail). The Kentucky River Regional Jail (KRRJ) is selected as the site for comparison group recruitment because it does not fall in the Mountain Comprehensive Care designated service region, and individuals residing in the KRRJ are comparable in demographics and other key variables of interest.

In the proposed evaluation, eligibility criteria used to select participants for the targeted MCCC grant-funded services in the Floyd County Detention Center and the Big Sandy Regional Detention Center will also be implemented in a comparison jail site. The Kentucky River Regional Jail (KRRJ) located in Hazard, Kentucky is not in the targeted service area for this MCCC project. KRRJ is comparable in size, characteristics of the offender population, and geographic location to the targeted facilities in Floyd County and Big Sandy. Following standardized screening based on grant eligibility criteria, the only anticipated difference between the experimental condition and the comparison condition is the opportunity to receive targeted services based on jail.

Following targeted screening, participants in the experimental (n=250) and comparison groups (n=250) will participate in baseline interviews focused on fatherhood, family relationships, and economic stability indicators, as well as factors which might impact these key outcomes including substance abuse and mental health. All participants in the local evaluation will also complete the post-test assessment at the conclusion of the courses (experimental group) or at a comparable time frame of 12 weeks for the comparison group. All evaluation participants will also be followed 6 months post-release from jail to complete an additional post-test assessment for the targeted instruments.

### **Study Population**

The MCCC estimates that during the first year a minimum of 50 participants will be served accounting for up to a 9-month planning period. It is estimated that 150 participants will be served annually in years 2-5, with a final total of 650 participants over 5 years. Of these participating individuals, 250 will be randomly selected (50 each year of the 5 year project) to be involved in the local evaluation. In addition, 250 comparison group participants will be recruited from a non-treatment site (jail). The 500 total participants recruited for the local evaluation will be incarcerated fathers. Participants for the local evaluation will be identified as eligible fathers who have been tried and convicted as an adult; within 3 to 9 months of release; are low-income; and may be an expectant father, a biological father, an adoptive father or a stepfather or who a person who is acknowledged as a father figure (e.g., grandfather) of a dependent child or young adult child up to 24 years of age, and interested in participation. The target population does not exclude individuals from participants because of age, race, ethnicity, sexual orientation, culture, literacy, disability, or language.

Based on data from the two targeted detention centers, 80% of all inmates are male and approximately 94% are parents. It is also anticipated that offenders will share similar characteristics to the targeted area including race (primarily White), chronic poverty, low educational attainment, high unemployment as well as 90% who have been arrested on alcohol or drug-related charges leading to family instability and separation. This population frequently faces not only the challenge of offender status but also substance use when trying to secure employment. Once enrolled in the evaluation, all participating clients will have access to the targeted ReFORM interventions. The local evaluation will enable analysis to focus on the unique contribution of enhancing parenting and relationship skills as well as job readiness and other employment and economic skills.

## **Subject Recruitment Methods and Privacy**

Recruitment efforts will target two groups of incarcerated fathers:

- 1) those who receive MCCC grant funded services (Floyd County Detention Center; Big Sandy Regional Jail, n=250); and
- 2) those who are incarcerated in jails not in the service delivery region for grant funded services (Kentucky River Regional Jail, n=250).

Participants in the treatment group will be informed about the local evaluation at treatment intake, and will be provided with an overview of the evaluation. If MCCC treatment participants are willing to be in the sampling frame for the local evaluation, they will sign the release of information form with the MCCC treatment coordinator. For the comparison group, the UK Program Coordinator will recruit participants from KRRJ once a month based on a randomized schedule. On each recruitment day, UK research staff will randomly select male offenders serving time in the jail from the daily census sheet to participate in the screening sessions. Jail personnel are not engaged in the research and not involved in the random selection of cases, and they will only providing access to the daily census sheet. UK research staff will randomly select 10-15 male participants residing in the jail on the day of screening. All male inmates will have an equal opportunity of being selected for the local evaluation, including minorities, as long as they are at least 18 years of age and not previously screened for the study.

Comparison group recruitment criteria will be matched to MCCC treatment participants including fathers who have been tried and convicted as an adult; within 3 to 9 months of release; are low-income; and may be an expectant father, a biological father, an adoptive father or a stepfather or a person who is acknowledged as a father figure (e.g., grandfather) of a dependent child or young adult child up to 24 years of age, and interested in participation. It is anticipated that approximately 5 comparison group participants will be recruited into the study each month in order to maintain a manageable number of participants for follow-up interviews.

# Advertising

N/A

#### **Informed Consent Process**

Names of interested and eligible treatment participants will be shared with the UK research staff after they sign a MCCC release of information. No research/evaluation activities will be initiated with the treatment participants until they meet with the UK research staff and sign informed consent. Comparison group participants who are interested in the study will be asked to participate in the screening session at the jail with the UK research coordinator. Potential participants in both conditions will be provided with informed consent prior to the collection of ANY data.

As part of the informed consent process, potential participants will be assured that:

- (a) Neither participation nor refusal to participate in a protocol will affect their legal parole status (if applicable);
- (b) No individual or identifiable data collected as part of a study protocol will be made available to any criminal justice authority including jail, parole, or community mandated treatment; and
- (c) If potential participants do NOT wish to participate, their parole or other legal status will not be affected. Potential participants who choose NOT to participate in the study protocol will not be identified in their records, and nonparticipation will NOT become a matter of official record in any file.

Informed consent procedures will cover participation in the screener (for the comparison group), baseline interview, and follow-up interviews so that participants are fully aware of all possible study procedures before making a decision about entering the study. Due to the sensitive nature of some of the questions asked in the interviews, confidentiality issues will be stressed during informed consent which will include a description of a federal Certificate of Confidentiality which provides an additional layer of human subject protection. Participants will also be assured that their screening results, study participation, and study data will not be made available to any representative of the criminal justice system. The research coordinator will keep detailed records on the number of interested participants who participate in the screening session and the number of refusals. Screening data will be examined as part of the implementation phase to examine characteristics of participants who enter the study compared to those who are not eligible. Because of the short time frame between baseline and follow-up interviews (approximately 12 weeks), consent procedures will not be repeated at each follow-up interview since no new procedures will be introduced. However, a follow-up script will be reviewed with The participant to remind him of the key elements of informed consent.

#### **Research Procedures**

To fulfill the requirements of the ACF funded grant, agency administrators and treatment staff are required to collect standardized performance measures. The evaluation PI will be given access to de-identified data through the ACF mandated nFORM data management system in order to assist the agency with data analysis for quarterly reports on:

1) program inputs (recruitment, enrollment, and characteristics of the client population);

- 2) program activities (quality assurance and monitoring, implementation challenges, and referrals to community agencies);
- 3) program outputs (enrollment, timing of client participation, program attendance, and overall program retention); and
- 4) program outcomes (changes in parenting behaviors, economic stability, relationships, personal development and well-being, and overall perceptions of the program).

These data are de-identified and required by the funding agency (ACF) to monitor program operations. This IRB application is focused primarily on the local evaluation. The nFORM data will only be used for the local evaluation with a signed release from the participant.

Potential local evaluation participants receiving targeted services at the Floyd County Detention Center or Big Sandy Regional jail will be asked about their interest in the local evaluation. If the participant is interested, he will be asked to sign a release of information to the evaluation team to access his nFORM information (specifically demographics and intake assessments which will be specified on the release). The UK research staff will work closely with MCCC project staff to identify individuals interested in the local evaluation.

Comparison group screening: Following random selection, the purpose of the screening session is to identify rural men who meet similar criteria as individuals receiving targeted MCCC services. The screening session (estimated 20 minutes) will be conducted between a trained study interviewer and the potential participants either in a face-to-face format or in a group setting, depending on the available jail accommodations. The session will include informed consent and an emphasis on the voluntary nature of study participation. Following consent, participants will be administered the ReFORM screening assessment (under development, will be forwarded for IRB approval prior to implementation). If the screener is administered in a group format, questions will be read aloud to participants and responses will be recorded confidentially on paper copies of the screener. Eligible participants will need to meet all of the specified study criteria to be invited to do a baseline interview.

<u>Data collection</u>: Potential comparison group participants meeting study eligibility criteria will complete a face-to-face baseline interview with the study interviewer the same day of the initial screening session, which is expected to last about 1 hour. Treatment group participants will also complete the required assessment interviews with the research staff after being identified as being interested in the local evaluation. The interviewer will be trained in the study protocol, as well as in jail policies and procedures. Interviews will be conducted in the jail visiting rooms which are large enough to provide a confidential face-to-face interview, and have been used to conduct interviews for other studies with offenders. While jail staff may monitor participant entry and exit into the visitation room, no jail staff will be present for the confidential interviews.

Data collection for the evaluation will include the initial Fatherhood Pre-test for Incarcerated Fathers, followed by an interview with the Evaluation Coordinator (in person, phone, or Wi-Fi audio) at 12 weeks post-intake (or completion of services), and again at 6 months post-release from jail. Participants will receive incentives for their time to complete data collection interviews.